CLINICAL TRIAL: NCT04489732
Title: Pilot Study of Mesenchymal Stromal Cells in Patients With Xerostomia After Radiation Therapy for Head and Neck Cancer
Brief Title: MSC in Patients With Xerostomia Post XRT in Head and Neck Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-1290; A533300 (Other: UW Madison); SMPH/HUMAN ONCOLOGY/HUMAN ONCO (Other: UW Madison); UW20025 (Other: UWCCC); NCI-2021-00070 (Registry Identifier: NCI CTRP); 1UG3DE030431-01 (NIH); Protocol Version 9/28/2023 (Other: UW Madison); Head & Neck SPORE (Other: Dr. Jacques Galipeau, MD)
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Results first posted 2024-02-23 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Xerostomia Following Radiotherapy

STUDY DESIGN:
Intervention Model Description: single-center, open-label, non-randomized, non-placebo controlled, single-group assignment, pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment with MSCs (Experimental): A single dose of MSCs injected into the submandibular glands of patients with radiation-induced xerostomia (primary objective)
  Following primary outcomes, a second injection of 10 (8 - 12) x 106 MSCs will be offered for injection into each participant's contralateral submandibular gland.
  Interventions: Biological: Autologous bone-marrow derived, interferon gamma stimulated mesenchymal stromal cells

INTERVENTIONS:
Biological: Autologous bone-marrow derived, interferon gamma stimulated mesenchymal stromal cells — Single dose, starting at
  * Dose Level 0: 10 (8-12) x 10^6 injected into one submandibular gland on Day 1
  Sub-study for second injection after primary objectives met, 10 (8 - 12) x 10^6 MSCs will be offered for injection into each participant's contralateral submandibular gland

SUMMARY:
This is a single center pilot study designed to determine the safety and tolerability of autologous bone marrow-derived Mesenchymal Stromal Cells (MSCs) in patients with xerostomia (dry mouth) after undergoing radiation therapy (XRT) for head and neck cancer (HNC). Up to 12 participants will be enrolled and can expect to be on study for up to 2 years.

DETAILED DESCRIPTION:
Following the completion of screening/baseline procedures, and written consent, eligible participants will undergo bone marrow aspirate in order to obtain MSCs.

The MSC Investigational Medicinal Product (IMP) (dose level 0, n=6, staggered) will be injected into one submandibular gland under local anesthesia, in the gland that received the lowest radiation dose. Patients with only one submandibular gland will be ineligible.

All participants will be called by a study coordinator 3 days (+/- 2 days) after injection to assess pain and will have a phone visit with a physician 1 week (+/- 2 days) after injection during which the investigator will assess pain and ask about the area of injection regarding redness and/or swelling. All participants will complete a pain diary with daily entries over the first month to record the occurrence and severity of pain using a 0-10 visual analog scale and occurrence and severity of other adverse events (e.g., redness, swelling, warmth, tenderness, rash, pruritis, nausea, vomiting, fatigue). Participants will also keep a log of all pain medications taken including both narcotic and non-narcotic medications (e.g. ibuprofen, acetaminophen, etc.) for the first month. Participants will complete 5 follow-up visits over the course of 24 months - at 1, 3, 6, 12, and 24 months following the intervention. Salivary collection for analysis as well as QoL surveys will be obtained at these visits.

Dose Reduction:

* If dose limiting toxicity (DLT) in less than or equal to 1 participant (n=6 participants, staggered at least 14 days), Dose Level 0 will be recommended as starting dose for subsequent trial.
* If DLT in greater than 1 participant, dose level -1 will be administered, staggered at least 14 days in n=6 participants.
* If DLT in this cohort is in less than or equal to 1 participant, Dose Level -1 will be recommended as starting dose for subsequent trial. If DLT in greater than or equal to 2 participants, study will be stopped.

Primary Objective

* To evaluate the safety and tolerability of MSCs for subjects with xerostomia after radiation therapy for HNC.

Secondary Objectives

* To evaluate the efficacy of MSCs for treatment of xerostomia and salivary hypofunction via quality-of-life (QoL) questionnaires, salivary amount, and salivary compositional analysis.
* To assess the imaging characteristics in HNC patients after MSC injection using ultrasound.
* To assess the feasibility of a future Phase 1 dose-escalation study.

Per Amendment Approved 4/14/23: Sub-study added, all enrolled participants will be offered injection of MSCs into the contralateral submandibular gland upon completion of the trial's primary objective (1 month of follow-up after injection of MSCs without any DLTs). The MSC IMP will be injected into the contralateral submandibular gland under local anesthesia.

Participants will complete 5 follow-up visits over the course of 24 months - at 1, 3, 6, 12, and 24 months following the contralateral injection. Salivary collection for analysis as well as QoL surveys will be obtained at all visits, except the 24 month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide informed consent
* Willing to comply with all study procedures and be available for the duration of the study
* Histological diagnosis of Head and Neck Cancer (HNC) and ≥ 2 years from completion of treatment for HNC, either clinically or radiologically No Evidence of Disease (NED), as assessed by ENT or Radiation Oncologist within 28 days of study registration
* Individuals at least 18 years of age and no older than 90 years of age
* Xerostomia defined as less than or equal to 80 percent of baseline (pre-radiation) salivary function per patient estimate
* Karnofsky performance status ≥ 70, patient eligible for bone marrow aspirate with wakeful anesthesia
* Radiographically confirmed bilateral submandibular glands
* Females of childbearing potential must agree to have a negative urine or serum pregnancy test within 7 days prior to bone marrow biopsy. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * has not undergone a hysterectomy or bilateral oophorectomy; or
  * has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* Women of childbearing potential in sexual relationships with men must have used an acceptable method of contraception for 30 days prior to study registration and agree to use an acceptable method of contraception until 4 weeks after completing study treatment. Males must agree to avoid impregnation of women during and for four weeks after completing study treatment through use of an acceptable method of contraception.

Note: Acceptable method of contraception includes, but is not limited to, barrier with additional spermicidal foam or jelly, intrauterine device, hormonal contraception (started at least 30 days prior to study enrollment), intercourse with men who underwent vasectomy)

Exclusion Criteria:

* History of sialolithiasis
* Patients with one submandibular gland
* History of autoimmune diseases affecting salivary glands, including Sjögren's syndrome, lupus, scleroderma, type I diabetes, sarcoidosis, and amyloidosis
* Chronic graft vs host disease
* Untreated oral candidiasis
* Use of anti-cholinergic medications (e.g. atropine, ipratropium, oxybutynin, scopolamine, solifenacin, tiotropium, etc…) while enrolled on study
* Malignancy within the past 2 years, except adequately treated stage I lung cancer, low risk prostate cancer that has been treated or is undergoing active surveillance, adequately treated non-melanoma skin cancer, adequately treated ductal carcinoma in situ (DCIS), or adequately treated stage I cervical cancer
* Expected life expectancy ≤ 6 months
* Lidocaine allergy
* Use of investigational drugs, biologics, or devices within 30 days prior to enrollment
* Women who are pregnant, lactating or planning on becoming pregnant during the study
* Not suitable for study participation due to other reasons at the discretion of the investigators

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2026-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Randall J Kimple, MD,PhD, Principal Investigator — University of Wisconsin, Madison; Jacques Galipeau, MD, Study Director — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blitzer GC, Glazer T, Burr A, Gustafson S, Ganz O, Meyers R, McDowell KA, Nickel KP, Mattison RJ, Weiss M, Chappell R, Rogus-Pulia NM, Galipeau J, Kimple RJ. Marrow-Derived Autologous Stromal Cells for the Restoration of Salivary Hypofunction (MARSH): A pilot, first-in-human study of interferon gamma-stimulated marrow mesenchymal stromal cells for treatment of radiation-induced xerostomia. Cytotherapy. 2023 Nov;25(11):1139-1144. doi: 10.1016/j.jcyt.2023.07.009. Epub 2023 Aug 15. PMID 37589639
- [Derived] Blitzer GC, Rogus-Pulia NM, Mattison RJ, Varghese T, Ganz O, Chappell R, Galipeau J, McDowell KA, Meyers RO, Glazer TA, Kimple RJ. Marrow-Derived Autologous Stromal Cells for the Restoration of Salivary Hypofunction (MARSH): Study protocol for a phase 1 dose-escalation trial of patients with xerostomia after radiation therapy for head and neck cancer: MARSH: Marrow-Derived Autologous Stromal Cells for the Restoration of Salivary Hypofunction. Cytotherapy. 2022 May;24(5):534-543. doi: 10.1016/j.jcyt.2021.11.003. Epub 2022 Feb 16. PMID 35183442

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at the UW Hospital and Clinics from February 2022 to September 2022.
Groups:
- Treatment With MSCs: A single dose of MSCs injected into the submandibular glands of patients with radiation-induced xerostomia
  Autologous bone-marrow derived, interferon gamma stimulated mesenchymal stromal cells: Single dose, starting at
  * Dose Level 0: 10 x 10^6 injected into one submandibular gland on Day 1
Period: Overall Study
Arm/Group | Treatment With MSCs
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment With MSCs
Number analyzed (Participants) | 6
Age, Customized [Count of Participants; unit: Participants]
  60-69 years | 2
  70-79 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Experiencing Dose Limiting Toxicity (DLT)
Description: Dose limiting toxicity is defined as: submandibular pain > 5 on a pain scale of 0-10 at 1-month after MSC injection OR any serious AE OR any of the selected toxicities listed per protocol within one-month post-injection.
Time Frame: up to 1 month post injection (up to 3 months from consent)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With MSCs
Number analyzed (Participants) | 6
Participants | 0

2. Secondary Outcome: Change in Saliva Production Rate
Description: Whole saliva production rates will be measured under unstimulated and stimulated saliva collection conditions.
Time Frame: baseline (up to 8 weeks before injection), 1, 3, 6, 12, and 24 months post-injection
Reporting Status: Not Posted

3. Secondary Outcome: Saliva Composition Analysis: Change in Salivary pH
Description: Salivary pH will be measured using a pH meter. The normal range of saliva pH is 6.2-7.6 .
Time Frame: baseline (up to 8 weeks before injection), 1, 3, 6, 12, and 24 months post-injection
Reporting Status: Not Posted

4. Secondary Outcome: Saliva Composition Analysis: Change in Total Protein Concentration in Saliva
Description: ELISA will be used to quantify total protein concentration in saliva. The normal range of total protein in saliva is 2-5 mg/mL.
Time Frame: baseline (up to 8 weeks before injection), 1, 3, 6, 12, and 24 months post-injection
Reporting Status: Not Posted

5. Secondary Outcome: Saliva Composition Analysis: Change in Amylase Concentration in Saliva
Description: The enzyme-linked immunosorbent assay (ELISA) will be used to quantify amylase concentration in saliva. The normal range of amylase concentration in saliva is 10-150 U/mL.
Time Frame: baseline (up to 8 weeks before injection), 1, 3, 6, 12, and 24 months post-injection
Reporting Status: Not Posted

6. Secondary Outcome: Saliva Composition Analysis: Change in Mucin Concentration in Saliva
Description: ELISA will be used to quantify mucin concentration in saliva.The normal range of mucin concentration in saliva is 1,000-3,000 ug/mL.
Time Frame: baseline (up to 8 weeks before injection), 1, 3, 6, 12, and 24 months post-injection
Reporting Status: Not Posted

7. Secondary Outcome: Change in The University of Michigan Xerostomia Related Quality of Life (XeQOL) Score
Description: The University of Michigan Xerostomia Related Quality of Life (XeQOL) scale is a validated patient-reported assessment 15 item scale with 4 domains: physical functioning, pain/discomfort, personal/psychologic functioning, and social functioning. Participants will answer the questions on a scale of 1-5 (not a all, a little, somewhat, quite a bit, very much) for every item. Higher scores represent greater degree of symptoms.
Time Frame: baseline (up to 8 weeks before injection), 1, 3, 6, 12, and 24 months post-injection
Reporting Status: Not Posted

8. Secondary Outcome: Change in The MD Anderson Dysphagia Index (MDADI) Score
Description: The MDADI is a 20-item questionnaire designed for evaluating the impact of dysphagia on the quality of life of patients with head and neck cancer. The MDADI score ranges from 20-100 with a lower scale representing worse dysphagia.
Time Frame: baseline(up to 8 weeks before injection), 1, 3, 6, 12, and 24 months post-injection
Reporting Status: Not Posted

9. Secondary Outcome: Change in Visual Analogue Scale (VAS) Xerostomia Score
Description: A Visual Analogue Scale questionnaire for subjective assessment of salivary dysfunction. The VAS xerostomia questionnaire is an 8-item questionnaire that provides a validated measure of the perception of dry mouth. Participants will be asked to mark their responses to each item by placing a vertical line on the 100-mm horizontal scale. The VAS ranges from 8-80 with a lower scale representing less dysphagia/symptoms
Time Frame: baseline (up to 8 weeks before injection), 1, 3, 6, 12, and 24 months post-injection
Reporting Status: Not Posted

10. Secondary Outcome: Change in Salivary Gland Size
Description: Salivary gland size measured by ultrasound imaging
Time Frame: baseline (up to 8 weeks before injection), 3, 6, and 12 months post-injection
Reporting Status: Not Posted

11. Secondary Outcome: Change in Salivary Gland Stiffness Measured by Shear Wave Velocity
Description: Salivary gland stiffness (fibrosis) will be measured by acoustic radiation force impulse imaging. Evaluators will be blinded to the time point of evaluation (pre- or post- MSC injection)
Time Frame: baseline (up to 8 weeks before injection), 3, 6, and 12 months post-injection
Reporting Status: Not Posted

12. Secondary Outcome: Participant Drop Out Rate
Description: Study feasibility will in part be measured by participant drop out rate.
Time Frame: up to 24 months post-injection (up to 26 months from consent)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Toxicities regardless of attribution were recorded through the 3 month post injection visit per protocol (up to 5 months from participant consent) for primary outcomes.
Description: Follow up for serious adverse events continues through 24 months post injection (up to 26 months from participant consent).
Arm/Group | Treatment With MSCs
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment With MSCs (N=6)
Injection Site reaction (pain) (General disorders) | 3
Vaccine site lymphadenopathy (General disorders) | 2
Lymphocyte decrease (Investigations) | 2
Bone pain (bone marrow aspiration) (Musculoskeletal and connective tissue disorders) | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Lymphedema (Vascular disorders) | 1
Platelet Count Decrease (Investigations) | 1
Cardiac Troponin 1 increase (Investigations) | 1
Anemia (Blood and lymphatic system disorders) | 1
Eosinophilia (Blood and lymphatic system disorders) | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-28): https://cdn.clinicaltrials.gov/large-docs/32/NCT04489732/Prot_SAP_001.pdf